CLINICAL TRIAL: NCT01228435
Title: A Phase II Study of IPI-204, A Novel Hsp90 Inhibitor in NSCLC Patients With ALK Translocations
Brief Title: IPI-504 in NSCLC Patients With ALK Translocations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-134; NCT01119495 (obsolete NCT alias)
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer; Stage IIIb Lung Cancer; Stage IV Lung Cancer
Keywords: NSCLC; IPI-504; ALK translocation; Hsp90 inhibitor
MeSH Terms: conditions — Lung Neoplasms | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALK-inhibitor naive (Experimental): No prior exposure to ALK-inhibitor
  Interventions: Drug: IPI-504
- ALK-inhibitor pre-treated (Experimental): Prior exposure to ALK inhibitor
  Interventions: Drug: IPI-504

INTERVENTIONS:
Drug: IPI-504 — Given intravenously twice weekly for 2 weeks followed by 10 day off treatment

SUMMARY:
IPI-504 blocks a protein that is in cancer cells and is also in normal cells. This protein is called Heat Shock Protein-90 (Hsp90). Hsp90 helps protect certain other proteins from being destroyed by cells. These proteins can mutate to give off signals that allow cancer cells to keep growing. By blocking the function of Hsp90, we hope that the cancer cell will block the mutated protein and cause the cancer cells to die. This drug have been used in other research studies and in the laboratory and information from those other research studies suggests that thsi drug may help to treat lung cancer with ALK mutations. In this research study, we are looking to see what effects IPI-504 has in patients with lung cancer who have an ALK mutation.

DETAILED DESCRIPTION:
* Participants will receive the study drug (IPI-504) twice weekly for two weeks followed by 10 days without study treatment. This 3-week period is called a cycle. Participants will receive a total of 4 doses per cycle. On the days the participant receives study drug, they will come to the clinic and be given the IPI-504 by being. Participants will continue to receive study drug for additional cycles as long as they are benefiting from it and do not experience any severe side effects.
* Participants will have CT scans to assess the size and location of their tumor. They may also have a PET scan or a combination of PET/CT scans. Imaging will be done at the beginning of treatment and every five to six weeks while on study to assess how the tumor is responding to IPI-504.
* The following tests and procedures will be done on the prior to the first dose of IPI-504: physical examination, vital signs, routine blood tests, EKGs, serum or urine pregnancy test (for women of child-bearing potential).
* After the first dose of IPI-504, the following tests and procedures will be done: EKGs, vital signs (pulse only).
* For all other visit days throughout the study, the following exams, tests and procedures will be done: physical examination, vital signs, blood tests, tumor imaging assessments, MRI of the brain (if applicable), review of medications and answer questions about any side effects or changes in health.
* After the final dose of study drug the following tests and procedures will be done within 30 days: physical examination, ECOG Performance status, blood tests, review of medications and answer questions about any side effects of changes in health.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed diagnosis of Stage IIIb (with malignant pleural or pericardial effusion), Stage IV, or recurrent NSCLC.
* Patients must have demonstrated ALK mutation
* There is no requirement for a minimum or maximum number of prior therapies, however, patients must have refused, be intolerant to or already received at least on standard systemic therapy for lung cancer
* Measureable disease by RECIST criteria. If a patient has received radiation therapy then measurable disease must be outside the radiation field.
* 18 years of age or older
* Life expectancy of at least 3 months
* ECOG performance status of 0-2
* Baseline studies for determining eligibility, except for ALK mutation status, must be completed within 30 days of first study dose.
* CT scan must be completed within 28 days prior to first study dose
* Women of child-bearing potential (WBCP) defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months must have a negative serum or urine pregnancy test within 2 weeks of first study dose
* All WCBP and all sexually active male patients must agree to use adequate methods of birth control throughout the study

Exclusion Criteria:

* Treatment for NSCLC with any approved or investigational product within 2 weeks of Cycle 1, Dose 1 for any small molecule therapy; within 4 weeks of Cycle 1, Dose 1 for any biologic or any conventional chemotherapy.
* Concurrent radiation therapy is not permitted
* Use of a medication or food that is clinically relevant CYP3A inhibitor or inducer within 2 weeks prior to Cycle 1, Dose 1
* Laboratory values as outlined in the protocol
* Baseline QT corrected using Fridericia's correction method (QTcf) > 470ms. Patients with left bundle branch block are eligible regardless of QTcf, as long as serum troponin is normal or undetectable
* Presence of active infection or systemic use of antibiotics within 72 hours of treatment
* Significant co-morbid condition or disease which in the judgment of the investigator would place the patient at undue risk or interfere with the study
* Women who are pregnant or lactating
* Previous treatment with 17-AAG, DMAG, or other known Hsp90 inhibitor
* Sinus bradycardia secondary to intrinsic conduction system disease. Patients with sinus bradycardia secondary to pharmacologic treatment may enroll if withdrawal of the treatment results in normalization of the resting heart rate to within normal limits
* Active keratitis or keratoconjunctivitis
* Alkaline phosphatase > 1.5 x ULN. Patients with bone metastases and an alkaline phosphatase level > 1/5 x ULN and less than or equal to 3 x ULN are eligible if they meet the criteria outlined in the protocol
* Prothrombin time (PT) and partial thromboplastin time (PTT) > 1.5 x ULN unless the patient is receiving warfarin. If the patient is receiving warfarin, the international normalized ratio must be within therapeutic range
* Patients with clinically active brain metastasis or an uncontrolled seizure disorder, ongoing spinal cord compression, or carcinomatous meningitis. Patients with clinically stable brain metastasis are eligible.
* Patients with prior hepatic resection or hepatic-directed therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V. Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the oncology clinic at Mass General from 6/10/10 to 9/26/11.
Pre-assignment Details: The study was closed to accrual after 3 patients were enrolled over a 1-year period. It was determined that there were too many competing protocols and completion of the study as designed was not feasible.
Groups:
- ALK-inhibitor Naive: Patients in this arm has no prior exposure to ALK-inhibitor and were treated with IPI-504 at 225 mg/m2 twice a week for 2 weeks followed by 10 days off therapy, cycles repeated every 21 days.
- ALK-inhibitor Pre-treated: Patients in this arm had prior exposure to an ALK inhibitor and were treated with IPI-504 at 225 mg/m2 twice a week for 2 weeks followed by 10 days off therapy, cycles repeated every 21 days.
Period: Overall Study
Arm/Group | ALK-inhibitor Naive | ALK-inhibitor Pre-treated
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALK-inhibitor Naive | ALK-inhibitor Pre-treated | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 | 67.5 (14.8) | 71.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The response rate was defined as the number of patients achieving a RECIST 1.0 defined response divided by the number of patients treated and was to be calculated separately for each arm. A response by RECIST criteria means that the pre-defined target lesions (sum of the longest diameters) had to decrease by 30% or more and this response needed to be confirmed on a second scan at least 4 weeks later.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- ALK-inhibitor Naive: Patients in this arm has no prior exposure to ALK-inhibitor and were treated with IPI-504 at 225mg/m2 twice a week for 2 weeks followed by 10 days off with cycles repeating every 21 days.
- ALK-inhibitor Pre-treated: Patients in this arm had received prior exposure to ALK-inhibitor and were treated with IPI-504 at 225mg/m2 twice a week for 2 weeks followed by 10 days off with cycles repeating every 21 days.
Arm/Group | ALK-inhibitor Naive | ALK-inhibitor Pre-treated
Number analyzed (Participants) | 1 | 2
participants | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Further document the safety of this regimen. Treatment-emergent adverse events will be summarized by MedDRA coding terms and separate tabulations will be produced for treatment-emergent adverse events, treatment-emergent serious adverse events, discontinuations due to adverse events, and treatment-emergent events of at least Grade 3 severity. A treatment-emergent adverse event is defined as an adverse event that was deemed to be related to the study intervention.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | ALK-inhibitor Naive | ALK-inhibitor Pre-treated
Number analyzed (Participants) | 1 | 2
participants
  Treatment-emergent adverse events | 0 | 0
  Treatment-emergent serious adverse events | 0 | 0
  discontinuations due to adverse events | 0 | 0
  treatment-emergent events ≥ grade 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | ALK-inhibitor Naive | ALK-inhibitor Pre-treated
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALK-inhibitor Naive (N=1) | ALK-inhibitor Pre-treated (N=2)
Fatigue (General disorders) | 1 | 0
Arthralgias (Musculoskeletal and connective tissue disorders) | 0 | 1
Elevated AST (Hepatobiliary disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was unable to accrue sufficient participants due to competing studies. Therefore, the study results are not sufficiently powered to draw any conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No